CLINICAL TRIAL: NCT01771354
Title: Clinical Study to Generate Exploratory Training Data Characterising Clinical Events, Physiological & Metabolic Responses, & Innate & Adaptive Immune Responses Following 1st & 3rd of 3 IM Immunisations With "Engerix B" HepB Vaccine or Placebo in Healthy Adults With no Pre-existing Immunity to HepB
Brief Title: Training Study to Characterise Biomarkers to the Engerix B Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: Innovative Medicines Initiative (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CRC305B
Record Dates: First submitted 2012-11-15; First posted 2013-01-18 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Volunteers; Identify; Biomarkers; Vaccine Safety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo
- Vaccine (Active Comparator): Engerix B vaccine
  Interventions: Biological: Engerix B Vaccine

INTERVENTIONS:
Biological: Engerix B Vaccine
  Arms: Vaccine
Biological: Placebo
  Arms: Placebo

SUMMARY:
It is thought that vaccines trigger innate inflammatory responses to induce antigenspecific adaptive immunity (the desired effect), but excessive inflammation may lead to serious inflammatory complications or unwanted side effects. Currently there is a lack of reliable biomarkers (a measurable biological response that predicts something) able to predict severe inflammation and this has resulted in the development of several vaccines being terminated and the withdrawal of some licensed vaccines which were associated with inflammatory complications.

This study is part of the BIOVACSAFE project which is a 5year €30M project funded by the Innovative Medicine Initiative. The project involves a series of clinical studies using licensed vaccines as benchmarks to generate clinical data on inflammation and identify biomarkers that can be used to predict acceptable reactogenicity. The target is to identify biomarkers that can predict the occurrence of beneficial and detrimental effects in response to a vaccine. Such biomarkers could be used in future vaccine development programs to optimize selection of vaccine candidates with a profile that will be unlikely to generate worrisome safety signals once they are in generalized use.

This study is one in a series of "training" studies which will each use different licensed vaccines that are prototypical representatives of a class of vaccine used in a particular target population. Twenty four subjects will be randomised into two groups to receive: A) Engerix B vaccine (n = 20), B) Saline placebo (n = 4). Following a screening visit, participants will undergo two immunisations at month 0 and month 6. Each immunisation will occur during a seven day residential visit which will include immunization and intensive monitoring of physiological (e.g. heart rate, oral temperature, blood pressure) metabolic and immune (innate and adaptive) parameters. Both residential visits will be followed up by four outpatient visits with further monitoring and blood samples.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18-45 years inclusive.
2. The subject is, in the opinion of the investigator, healthy on the basis of medical history, vital signs, & the results of routine laboratory tests with no active disease process that could interfere with the study endpoints.
3. Body Mass Index ≥18.5 & <29.5
4. The subject is able to read & understand the Informed Consent Form (ICF), & understand study procedures.
5. The subject has signed the ICF.
6. The subject has not previously received a vaccine for Hepatitis B or contracted hepatitis B infection.
7. The subject is seronegative to Hepatitis B as confirmed at screening by assessments of sAb, sAg, & cAb.
8. Available for followup for the duration of the study.
9. Agree to abstain from donating blood during & for three months after the end of their participation in the study, or longer if necessary.
10. If heterosexually active female, willing to use an effective method of contraception with partner from 30 days prior to, & 3 months after, vaccination. Willing to undergo urine pregnancy tests prior to vaccination & blood pregnancy test at screening & final follow up.
11. The subject has venous access sufficient to allow blood sampling as per the protocol.

Exclusion Criteria:

1. Significant dietary restrictions (e.g. vegan, lactose intolerant, but vegetarian acceptable) or life-threatening food allergies (e.g. anaphylaxis related nut allergies).
2. Pregnant or lactating at any point during the study from screening to final follow up.
3. Known hypersensitivity to any component of the vaccine (excipients: sodium chloride, disodium phosphate dehydrate, sodium dihydrogen phosphate; Hepatitis B antigen produced in yeast cells) or subjects who have exhibited hypersensitivity following previous Engerix B administration; or known hypersensitivity to any other hepatitis B vaccine.
4. Presence of primary or acquired immunodeficiency states with a total lymphocyte count less than 1,200 per mm3 or presenting other evidence of lack of cellular immune competence e.g. leukaemias, lymphomas, blood dyscrasias, or patients receiving immunosuppressive therapy (including regular use of oral, inhaled, topical or parenteral corticosteroids).
5. Use of any immune suppressing or immunomodulating drugs within 6 months of Visit 1 (screening).
6. Regular use of nonsteroidal antiinflammatory drugs (by any route of administration including topical) within 6 months of Visit 1 (screening) considered by the study physician as likely to interfere with immune responses.
7. Receipt of a vaccine within 30 days of visit 2, or requirement to receive another vaccine within the study period.
8. Presence of an acute severe febrile illness at time of immunisation.
9. History of alcohol, narcotic, benzodiazepine, or other substance abuse or dependence within the 12 months preceding Visit 1.
10. Currently participating in another clinical trial with an investigational or noninvestigational drug or device, or has participated in a clinical trial within the 3 months preceding Visit 1.
11. Any condition that, in the investigator's opinion, compromises the subject's ability to meet protocol requirements or to complete the study.
12. Receipt of blood products or immunoglobin, or blood donation, within 3 months of screening.
13. Unable to read & speak English to a fluency level adequate for the full comprehension of procedures required in participation & consent.
14. An average weekly alcohol intake that exceeds 14 or 21 units per week for females & males, respectively, or unwilling to stop alcohol consumption for each treatment period during the study.
15. Currently smokes in excess of 5 cigarettes/day or equivalent use of tobacco (within the last 6 months of screening), or subjects unwilling to refrain from smoking or are unable to abide by Surrey CRC restrictions.
16. Consumes excessive amounts, defined as greater than 4 servings of coffee, tea, cola, or other caffeinated beverages/food per day.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline values of global gene expression in whole blood. | Visits 1 (Day -28 to -2), 2 (Day -1 to +5) , 3 (Day 7), 4 Day 14), 5 (Day 21), 6 (Day 28), 7 (Day 168 to 173), 8 (Day 175), 9 (Day 182), 10 (day 189), 11 (Day 196).

OTHER OUTCOMES:
Proportion of subjects experiencing vaccine-related clinical events following administration of vaccine. | Visits 2 (Day -1 to +5) , 3 (Day 7), 4 Day 14), 5 (Day 21), 6 (Day 28), 7 (Day 168 to 173), 8 (Day 175), 9 (Day 182), 10 (day 189), 11 (Day 196).

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, Professor, Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Surrey CRC, Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Weiner J, Lewis DJM, Maertzdorf J, Mollenkopf HJ, Bodinham C, Pizzoferro K, Linley C, Greenwood A, Mantovani A, Bottazzi B, Denoel P, Leroux-Roels G, Kester KE, Jonsdottir I, van den Berg R, Kaufmann SHE, Del Giudice G. Characterization of potential biomarkers of reactogenicity of licensed antiviral vaccines: randomized controlled clinical trials conducted by the BIOVACSAFE consortium. Sci Rep. 2019 Dec 30;9(1):20362. doi: 10.1038/s41598-019-56994-8. PMID 31889148
- See also: BIOVACSAFE — http://www.biovacsafe.eu/